CLINICAL TRIAL: NCT01657643
Title: Effect of Lactobacillus Rhamnosus LGG® and Bifidobacterium Animalis Ssp Lactis BB-12® on Health-related Quality of Life in College Students With Upper Respiratory Infections
Brief Title: Effect of Probiotics on Health-related Quality of Life in College Students With Upper Respiratory Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: Chr Hansen A/S (Unknown)
Responsible Party: Principal Investigator, SHRP nutritional sciences, Tracey J. Smith, Doctoral Student, Rutgers, The State University of New Jersey
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 0120100395
Record Dates: First submitted 2012-07-28; First posted 2012-08-06 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Upper Respiratory Infection
Keywords: Health related quality of life; Functional Status
MeSH Terms: conditions — Respiratory Tract Infections | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Every day for 12 weeks, subjects are asked to eat 5 grams of a placebo (strawberry-flavored candy powder)
  Interventions: Dietary Supplement: placebo
- Probiotics (Experimental): Every day for 12 weeks, subjects are asked to eat 5 grams of a strawberry-flavored candy that contains probiotics [daily dose minimum of 1 billion CFU of each Lactobacillus rhamnosus LGG® (LGG®), and Bifidobacterium animalis ssp lactis BB-12® (BB-12®)]
  Interventions: Dietary Supplement: Probiotics

INTERVENTIONS:
Dietary Supplement: Probiotics
  Other Names: Lactobacillus rhamnosus LGG® (LGG®); Bifidobacterium animalis ssp lactis BB-12® (BB-12®)
  Arms: Probiotics
Dietary Supplement: placebo
  Arms: Placebo

SUMMARY:
The main purpose of the study is to find out if probiotics (healthy bacteria found in yogurt) can improve the health-related quality of life (HRQL) during upper respiratory infections (like the common cold) in college students living in residence hall on-campus at Framingham State University (Framingham, MA) who are randomized to receive a probiotic or placebo candy daily for 12 weeks. HRQL is a subjective measure, defined as the aspects of quality of life (i.e., one's satisfaction with their life) that related specifically to a person's health (for example, ability to carry out normal daily activities). The investigators hypothesize that HRQL during URIs will be significantly higher in the probiotic groups compared to the placebo group. The proposed study will also seek to address the following secondary objectives: missed school and work days due to a upper respiratory infection.

ELIGIBILITY:
Inclusion Criteria:

1. Student at Framingham State University (Framingham, MA)
2. Live in on-campus housing

Exclusion Criteria:

1. their driver's license or state identification card indicated that they were under 18 years of age or over 25 years of age;
2. they experienced chronic perennial allergies (such as, allergies to dust or 3) they were pregnant

4) they had been diagnosed with medical conditions affecting immune function (for example, asthma, chronic fatigue syndrome and human immunodeficiency virus) 5) they had acute pancreatitis, were undergoing treatment for cancer; or, were taking immunosuppressive drugs for an autoimmune disease or post-transplant.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 231 (Actual)
Dates: Start 2011-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life | 12 weeks
  Subjects are asked to complete a questionnaire every day for 12 weeks that inquires about any common cold symptoms that they may be experiencing, severity of the symptoms, and how the symptoms interfere with their daily activities. Health-related quality of life is operationalized by total score on the questionnaire.

SECONDARY OUTCOMES:
Missed work days | Once per week over the course of 12 weeks
  Once per week, for 12 weeks, subjects are asked to complete a questionnaire that inquires about missed work days.

OTHER OUTCOMES:
Missed school days | Once per week over the course of 12 weeks
  Once per week, for 12 weeks, subjects are asked to complete a questionnaire that inquires about missed school days.

CONTACTS AND LOCATIONS:
Overall Officials: Tracey J Smith, PhD, Principal Investigator — University of Medicine and Dentistry of New Jersey
Locations (1):
- Framingham State University, Framingham, Massachusetts, United States